CLINICAL TRIAL: NCT04096794
Title: Chinese Alliance for Type 1 Diabetes Multi-center Collaborative Research
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Professor,Institute of Metabolism and Endocrinology, The Second Xiangya Hospital and the Diabetes Center, Key Laboratory of Diabetes Immunology, Ministry of Education, Central South University, National Clinical Research Center for Metabolic Diseases., Second Xiangya Hospital of Central South University
Other Study IDs: CAT1D2019CS0011
Record Dates: First submitted 2019-09-02; First posted 2019-09-20 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The China Alliance for Type 1 Diabetes (CAT1D) is committed to exploring and implementing the model of graded diagnosis and treatment of type 1 diabetes and comprehensive management of outpatient service, carrying out a series of educational activities for patients, and cooperating in the development of multi-center prospective clinical research on type 1 diabetes.

DETAILED DESCRIPTION:
1. Through the CAT1D, expand the cohort construction of type 1 diabetes patients and first-level relatives in China, establish the electronic information database of type 1 diabetes, and lay a foundation for obtaining the research data of type 1 diabetes in China.
2. observe and study the occurrence and development rules of acute and chronic complications of type 1 diabetes in China, analyze the influencing factors, and provide intervention means for reducing acute complications and preventing chronic complications.
3. Through the established management platform and structured education system, verify and promote the comprehensive management mode based on structured education, and build a standard treatment plan and process based on evidence-based science and suitable for Chinese people and medical background.
4. By using mobile health (mHealth) and Artificial Intelligence (AI) technologies, a new mode of intelligent structured education is established, which provides a new way to explore the individualized education management mode and improve the outcome of chronic diseases through modern technology.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Type 1 Diabetes according to the 1999 World Health Organization report
* Written informed consent from the patient or family representative;
* Individuals who own smartphone and are capable of using wechat or apps

Exclusion Criteria:

* Non-t1dm patients with autoimmune polyendocrine adenopathy syndrome (APS) are the first disease
* With mental disorders
* Have any other condition or disease that may hamper from compliance with the protocol or complication of the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: type 1 diabetes patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
changes in serum hemoglobin A1c level | Baseline and every up to 12 weeks afterwards
  A1c reflects the average blood glucose level in the past 3 months.

SECONDARY OUTCOMES:
changes in Time in range (TIR) | Baseline and every up to 12 weeks afterwards
  TIR measures the time where the blood glucose remains within the proposed target range.
C-peptide | Baseline and every up to 12 weeks afterwards
  C-peptide are measured before and 2-hour after a mixed meal tolerance test at each follow-up of this study
Change in titer of autoantibodies | Baseline and every up to 12 weeks afterwards
Fasting blood glucose | Baseline and every up to 12 weeks afterwards
  the blood sugar level after fasting for eight hours
Systolic blood pressure | Baseline and every up to 12 weeks afterwards
  Systolic blood pressure
Diastolic blood pressure | Baseline and every up to 12 weeks afterwards
  Diastolic blood pressure
Change in lipid profiles | Baseline and every up to 12 weeks afterwards
  Including triglyceride, total cholesterol, HDL-cholesterol and LDL-cholesterol
Height in meters | Baseline and every up to 12 weeks afterwards
  Height in meters will be measured
Weight in kilograms | Baseline and every every up to 12 weeks afterwards
  Weight in kilograms will be measured
Stool samples | Baseline and every up to 12 weeks afterwards
Adverse effects | Baseline and every up to 12 weeks afterwards
  Adverse effects are recorded at each time-point of the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided